CLINICAL TRIAL: NCT06510855
Title: DurAVR™ THV System: European Early Feasibility Study
Brief Title: DurAVR™ THV EU-EFS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anteris Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: SP0082
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Symptomatic Aortic Stenosis; Severe Aortic Valve Stenosis; Aortic Valve Calcification; Aortic Valve Failure; Aortic Valve Disease
Keywords: Transcatheter Aortic Valve Implantation (TAVI); Transcatheter Aortic Valve Replacement (TAVR); Transcatheter Valve; Valve-in-Valve; Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve, Calcification of; Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Severe Aortic Stenosis (sAS) Cohort (Experimental): Subjects with symptomatic severe native aortic stenosis with a Heart Team determination of eligibility for delivery of the DurAVR™ THV prosthesis.
  Interventions: Device: DurAVR™ THV System
- Failed Surgical Aortic Bioprosthetic Valve (FAV) Cohort (Experimental): Subjects with severe degeneration of surgically implanted aortic bioprosthetic valves with a Heart Team determination of eligibility for delivery of the DurAVR™ THV prosthesis.
  Interventions: Device: DurAVR™ THV System

INTERVENTIONS:
Device: DurAVR™ THV System — DurAVR™ THV System - Transcatheter Aortic Valve Implantation (TAVI) Procedure

SUMMARY:
A prospective, non-randomized, single-arm, multi-center study designed to evaluate the safety and feasibility of DurAVR™ THV System in the treatment of subjects with symptomatic severe native aortic stenosis or failed surgical aortic bioprosthetic valves.

DETAILED DESCRIPTION:
The DurAVR™ THV System is a novel balloon-expandable single-piece transcatheter aortic valve.

The study will enroll up to 40 subjects with severe, symptomatic native aortic stenosis or with severe degeneration of surgically implanted aortic bioprosthetic valves, with a Heart Team determination of eligibility for delivery of the DurAVR™ THV prosthesis.

Subjects will be consented for follow-up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic, severe native aortic stenosis or severe degeneration of surgically implanted aortic bioprosthetic valve in subjects 18 years or older.
2. Requires aortic valve replacement and is indicated for TAVR as determined by the Heart Team
3. Eligible for transfemoral delivery of the DurAVR™ THV
4. Anatomy appropriate to accommodate safe placement of DurAVR™ THV
5. Understands the study requirements and the treatment procedures and provides written informed consent
6. Subject agrees to complete all required scheduled follow-up visits.

Exclusion Criteria:

1. Anatomy precluding safe placement of DurAVR™ THV
2. Pre-existing prosthetic mitral or tricuspid valve
3. Unicuspid, bicuspid or non-calcified aortic valve
4. Severe mitral or severe tricuspid regurgitation requiring intervention
5. Moderate to severe mitral stenosis
6. Hypertrophic obstructive cardiomyopathy
7. Echocardiographic evidence of intracardiac mass, thrombus or vegetation requiring treatment
8. Evidence of an acute myocardial infarction ≤ 30 days before the intended treatment
9. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to the index procedure
10. Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA)
11. End-stage renal disease requiring chronic dialysis or creatinine clearance < 20 cc/min
12. GI bleeding within the past 3 months
13. Ongoing sepsis (including active endocarditis) or endocarditis in the last 3 months
14. Life expectancy < 12 months due to associated non-cardiac co-morbid conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality or disabling stroke | 30 Days
  Mortality would be reported as rate of death/mortality at 30 days. Disabling stroke would be reported according to VARC-3 Guidelines

SECONDARY OUTCOMES:
All-cause mortality | 30 Days
  Mortality would be reported as rate of death/mortality at 30 days.
Disabling stroke | 30 Days
  Disabling stroke would be reported according to VARC-3 Guidelines
Life-threatening bleeding | 30 Days
  Life-threatening bleeding according to VARC-3 Guidelines
Major vascular, access-related, or cardiac structural complication | 30 Days
  Major vascular, access-related, or cardiac structural complication according to VARC-3 Guidelines
Acute kidney injury stage 3 or 4 | 30 Days
  AKI according to VARC-3 Guidelines
Moderate or severe aortic regurgitation | 30 Days
  Aortic regurgitation according to VARC-3 Guidelines
New permanent pacemaker due to procedure related conduction abnormalities | 30 Days
  Rate of pacemaker interventions in subjects experiencing conduction abnormalities (sAS cohort only)
Surgery or intervention related to the device, including aortic valve reintervention | 30 Days
  Device related interventions

IPD SHARING:
Plan to Share IPD: No